CLINICAL TRIAL: NCT06928389
Title: A Randomized, Double-blind, Multicenter Phase 3 Clinical Trial of Ivonescimab Versus Placebo, Combined With Docetaxel in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) That Has Progressed on or After PD-(L)1 Inhibitor-based Therapy
Brief Title: Ivonescimab in Combination With Docetaxel in Advanced Non-Small Cell Lung Cancer
Acronym: NSCLC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK112-305 (HARMONi-8A)
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivonescimab and docetaxel (Experimental)
  Interventions: Drug: Ivonescimab, docetaxel
- Placebo and docetaxel (Active Comparator)
  Interventions: Drug: Placebo, docetaxel

INTERVENTIONS:
Drug: Ivonescimab, docetaxel — Patients will receive ivonescimab and docetaxel as an IV injection
  Other Names: AK112, docetaxel
  Arms: Ivonescimab and docetaxel
Drug: Placebo, docetaxel — Patients will receive placebo and docetaxel as an IV injection
  Arms: Placebo and docetaxel

SUMMARY:
This is a Phase 3 Randomized, double-blind, Multicenter Study of Ivonescimab Combined with Docetaxel Versus Placebo Combined with Docetaxel in Patients with Locally advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) that has progressed on or after PD-(L)1 inhibitor-based therapy. The purpose of this study is to evaluate the efficacy and safety of ivonescimab versus placebo, combined with docetaxel in patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Age ≥ 18 years old and ≤ 75 years old at the time of randomization.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected life expectancy of at least 3 months.
* Histologically or cytologically confirmed diagnosis of NSCLC.
* Locally advanced or metastatic NSCLC (American Joint Committee on Cancer [AJCC] 8th edition).
* Previously received systemic platinum-based chemotherapy and PD-1/L1 inhibitors.
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Adequate organ function.

Exclusion Criteria:

* Histologic or cytopathologic evidence of the presence of small cell lung carcinoma.
* Other malignancies within 3 years prior to randomization.
* Known actionable genomic alterations.
* Prior administration of any immunotherapy targeting immune mechanisms other than PD-1/PD-L1 inhibitors.
* Previous treatment with docetaxel.
* History of severe bleeding tendency or coagulation dysfunction.
* Active autoimmune disease requiring systemic therapy within 2 years prior to randomization.
* History of myocarditis, cardiomyopathy, and malignant arrhythmia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | approximately 5 years
  Overall Survival (OS) in the FAS population

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | approximately 3 years
  Progression Free Survival (PFS) assessed by investigator based on RECIST V1.1
Adverse Event (AE) | From the patient signs the ICF to 30 days (AE) and 90 days (SAE) after the last dose of study treatment or initiation of other anticancer therapy, whichever occurs first
  Incidence and severity of adverse events (AEs) and clinically significant abnormal laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai East Hospital